CLINICAL TRIAL: NCT03624140
Title: Hemoglobin Monitoring During High Bleeding Risk Surgery in Pediatric Patients: Equivalence Study of Hemoglobin Transcutaneous Saturation and Hemocue With Total Serum Hemoglobin
Brief Title: A Comparison of Three Methods of Hemoglobin Monitoring in Pediatric Patients
Acronym: HEMOPED2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-A01379-46
Record Dates: First submitted 2018-08-07; First posted 2018-08-09 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Child
Keywords: major pediatric surgery; hemoglobin measurement

STUDY DESIGN:
Intervention Model Description: Blood measurement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemoglobin monitoring (Experimental): 3 different techniques will be used for hemoglobine monitoring : hemocue, pulse co-oxymeter (SpHb) and blood measurement
  Interventions: Device: blood measurement; Device: pulse co-oxymeter (SpHb); Device: hemoCue

INTERVENTIONS:
Device: blood measurement — Hemoglobin measurement
Device: pulse co-oxymeter (SpHb) — non invasive method of hemoglobin measurement
Device: hemoCue — non invasive method of hemoglobin measurement

SUMMARY:
Investigators compare the accuracy of the SpHb and hemocue with blood Hb levels

DETAILED DESCRIPTION:
The goal of the study is to compare 3 methods of hemoglobin measurement in pediatric patients undergoing major surgery. During general anesthesia investigators will measure and compare at different periods of time blood hemoglobin levels obtained from a radial artery catheter with 2 non invasive methods of measurement using hemocue and SpHb

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients scheduled for surgery under general anesthesia
* Arterial catheter necessary in the anesthetic protocol
* BMI<30
* Written consent of holders of parental authority
* No opposition of children

Exclusion Criteria:

- Hemoglobine disease

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 195 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
level of hemoglobin using 3 different techniques at the time of transfusion decision | within the day of surgery
  comparison of blood hemoglobin obtained by arterial samples with 2 non invasive methods of measurement using hemocue and SpHb